CLINICAL TRIAL: NCT03248895
Title: Evaluation of a Mobile Direct Observation Therapy (DOT) Approach in Children and Young People With Asthma. Pilot Study
Brief Title: Evaluation of a Mobile Direct Observation Therapy (DOT) Approach in Children and Young People With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, James McElnay, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUB B14/39
Record Dates: First submitted 2017-08-03; First posted 2017-08-15 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Asthma in Children
Keywords: Inhaler assessment; Direct observation of therapy

STUDY DESIGN:
Intervention Model Description: A randomised intervention trial will be used. Participants will be randomised to either an immediate (I-med) or a delayed (D-med) intervention. Randomisation will be restricted based on two factors including age and patient gender.
  Both subject groups will receive standard-of-practice asthma education and management in the Asthma Clinic prior to study enrolment. Participants allocated to the I-med group will take part in the mobile technology DOT intervention for the first 6 weeks. Outcomes will be evaluated at the start (week 0) and end of the 6 week intervention period and during clinic visits at weeks 12 and 18 for follow-up. Those participants allocated to the D-med group will have the DOT intervention started after a 6 week "intervention-free" interval with usual Asthma Clinic care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (I-med) (Active Comparator): Participants allocated to the I-med group will take part in the mobile DOT intervention for the first 6 weeks. Outcomes will be evaluated at the start (week 0) and end of the 6 week intervention period and during clinic visits at weeks 12 and 18 for follow-up
  Interventions: Device: Mobile Direct Observation of Therapy (MDOT)
- Delayed (D-med) (Active Comparator): Those participants allocated to the D-med group will have the DOT intervention started after a 6 week "intervention-free" interval with usual Asthma Clinic care. Outcomes in the D-med group will be assessed at baseline (week 0), week 6 (intervention start), week 12 (end of intervention), and at weeks 18 and 24 for follow-up.
  Interventions: Device: Mobile Direct Observation of Therapy (MDOT)

INTERVENTIONS:
Device: Mobile Direct Observation of Therapy (MDOT) — Patients who are enrolled in the study will be randomised into two groups (I-med or D-med) to receive Mobile Direct Observation of Therapy (MDOT). Participants or parents/guardians of participants will be asked to capture a DOT video twice daily (morning and evening) on their mobile devices of ICS use by the patient. In the I-med group, participants will be asked to upload daily video recordings via the internet to a repository for a 6 week period at the start of the study. Participants in the D-med group will be free from DOT for the first 6 weeks of the study and will be asked to carry out their usual therapy management. After that, DOT as described above will be applied for the next 6 weeks.

SUMMARY:
Mobilte Direct Observation Therapy (MDOT) is a technology has the potential to be a cost effective approach to direct observation of therapy administration, the latter being one of the most accurate methods of evaluating adherence. Use to date, as confirmed by the rapid systematic review, has been limited mainly to TB and sickle cell disease and there have been no published reports on the use of MDOT to monitor inhaled therapy. Due to the increasing incidence of childhood asthma worldwide, there is a need for new innovative approaches to support children and their parents with asthma management, especially since national and international guidelines have advised healthcare providers to periodically assess inhaler use as part of asthma management.

DETAILED DESCRIPTION:
Asthma is the most common chronic disease in childhood. It is defined as a chronic inflammatory disorder of the airways in which many cells and cellular elements promote airway obstruction and hyper-responsiveness (GINA, 2012). According to the World Health Organization (WHO, 2014), asthma is estimated to affect approximately 253 million people worldwide. Despite advances in biological and pathological research, the prevalence of asthma in children has significantly increased over the past decade (Massingham et al., 2014).

Moreover, the economic burden of asthma is increasing. In the US, it is estimated that the yearly cost of asthma in children and adults is around $1.48 billion (Price et al., 2013). A decade ago, the total annual asthma expenditure in the UK was determined to be £752.6 million with 8% of costs associated with hospital admission, 13% attributable to general practitioner consultations and 79% due to prescription costs (Gupta et al., 2004).

The British Thoracic Society (BTS/SIGN, 2012) and Global Initiative for Asthma (GINA, 2012) guidelines provide the background definitions for three broad categories of asthma control. They include controlled (no nocturnal wakening, infrequent short acting beta 2 agonist (SABA) use e.g. < 2 puffs/week, occasional mild symptoms e.g. with exercise and no exacerbations in last 3 months), partially controlled (nocturnal wakening < 3 nights/week, SABA use e.g. < 4 puffs/day, mild limitation in exercise tolerance due to asthma, and 2 or fewer mild exacerbations in the previous 3 months) or uncontrolled (nocturnal wakening 4-7 nights/week, SABA use e.g. > 5 puffs/day, limitation in exercise tolerance due to asthma and or significant asthma exacerbations requiring oral steroid, Emergency Department attendance or hospital admission in the previous 3 months). Children who present with partially controlled or uncontrolled asthma can be divided into difficult to treat asthma (DTA) and true severe therapy resistant asthma (STRA) after careful investigation (Hedlin et al., 2012). DTA occurs when asthma is uncontrolled but the impact of concomitant disorders and the basics of asthma care (inhaler technique and adherence) have not been adequately resolved.

Many children with asthma can achieve symptom and disease control by using inhaled corticosteroid (ICS) therapy combined with a long acting B2 agonist (LABA) and/or a leukotriene receptor antagonist (LTRA) (International ERS/ATS guideline, 2014). However, a number of children with asthma experience frequent symptoms despite being prescribed high dose ICS (Nagakumar and Thomas, 2013; Hedlin et al., 2014).

Drug delivery by inhalation of various medications is the most common treatment approach for asthma in all patient populations. Inhalation therapy offers rapid onset and improved efficacy compared to systemic drug delivery (Bisgaard, 1997). While ICS therapy is well accepted as the foundation of optimal therapy for most asthma patients, efficacy of the therapy depends on drug being delivered correctly into the lungs and taken on a regular basis as a preventer therapy (Machira et al., 2011).

It has been suggested that good inhaler technique is an essential aspect of optimal asthma management. Education on inhaler technique has been shown to improve self- management and adherence to asthma therapy. Evidence is available demonstrating that asthma outcomes correlate with proper inhaler technique and that periodically assessing this treatment aspect has a positive impact on asthma control (Bryant et al., 2013; AL-Jahdali et al., 2013). Moreover, early and repeated tailored education and follow-up assessment can result in sustained good inhaler technique (Klot et al., 2011). However, many asthma clinics treating children are unable to effectively evaluate these important patient treatment variables.

Adherence to pharmacotherapy is also considered an important basic tenet of asthma management. Adherence can simply be defined as the extent to which a patient follows the instructions of the prescriber (Osterberg and Blaschke, 2005). While inhaled therapy technique is an essential feature of asthma pharmacotherapy, some patients with good technique may have poor inhaler adherence. Available data suggest the average medication adherence to ICS in children is only approximately 50% (Fish et al., 2001; Osterberg and Blaschke, 2005).

It is known that adherence to ICS in children is a complicated matter influenced by diverse issues including socioeconomic factors, parents' beliefs about asthma and asthma medications, and poor patient-doctor communication (Osterberg and Blaschke, 2005; Armstrong et al., 2014). In addition, parent/guardian health issues such as depression or substance abuse may negatively affect adherence in young children as a result of the parent/guardian's failure to remind, or assist the child in the use of their medication (Brackis-Cott et al., 2003). Non-adherence to medication can have various negative patient consequences such as more frequent clinic visits, disease exacerbations, hospital admissions, and increased cost of care (AL-Jahdali et al., 2013). Indeed, a recent review of childhood asthma deaths in SE England showed that medication non-adherence was a contributing factor in more than 50% of cases, including patients with milder disease (Anagnostou et al.,2012) Despite being an area of active research, many interventions such as isolated educational efforts are ineffective in improving adherence (Drotar and Bonner, 2009). In a qualitative study in the primary care setting, asthmatic children of parents who expressed medication beliefs of a high concern-low need pattern had poor outcomes. Researchers subsequently showed that these beliefs could be modified by repeated tailored education and close follow-up, to result in high medication adherence. They concluded that "it is not the education per se, but rather the intensity, quality and frequency of education about self-management and follow-up that help to improve adherence" (Klot et al., 2011). A multicentre clinical trial in the USA was designed to determine what medication was best to add in children with severe asthma already taking ICS and LABA. However,the trial was cut short due to an inability to recruit an adequate number of children. Patient improvement while under close supervision during the run in period was the main reason for the lack of patient recruitment. (Strunk et al., 2008) Different methods used to assess patient adherence to prescribed therapy have resulted in variable outcomes. Adherence can be measured by collecting data from patients or their parent/guardians, pharmacy dispensing records, electronic monitoring devices, or patient observation (Osterberg and Blaschke, 2005). Since the approaches have produced variable results, it can be concluded that presently there is no preferred method to effectively measure or improve medication adherence in asthma (Sumino and Cabana, 2013).

Direct observation therapy (DOT) is recommended by the WHO to promote adherence in the management of tuberculosis (TB) and this approach was adopted in 187 countries by 2005 (WHO, 2010). DOT allows assessment of correctly taking and completing therapy, but also can be valuable to promote adherence to medication use. DOT involves a healthcare professional observing patients taking their medication at home or in the clinic (Dosumu, 2001; Otu, 2013). The DOT approach to TB management has been utilised successfully in different countries as this approach has been shown to enhance medication adherence, improve outcomes including microbiologic success, and decrease acquired drug resistance to therapy (Favorov et al., 2012; Walley et al., 2001; Pasipanodya and Gumbo, 2013).

While data exist to show that observation of inhaler technique can positively affect asthma management, there are no published studies using a DOT approach as a means to improve medication adherence. However, it has been suggested that using DOT with nurses directly observing asthmatic children's inhaler technique and adherence, for example at school or home, would be very resource intensive and likely not feasible for continued use (Otu, 2013).

In recent years, there has been widespread use of mobile smartphone and computer devices within the healthcare environment. A recent survey of teenagers and caregivers in urban paediatric practices showed that 84% of respondents were smartphone owners, a finding that was independent of age group, gender, ethnicity, and socioeconomic status (Singh et al., 2014). DeMaio et al. (2001) conducted a pilot study that compared videophone telemedicine (V-DOT) to standard DOT (S-DOT) in the treatment of TB. In the videophone group, patients took videos of medication administration that were provided to clinicians involved in their management. The adherence rate was 95% for V-DOT compared to 97.5 % for S-DOT, but personnel time was decreased by 288 hours with V-DOT in only 6 patients. Similarly, a telehealth videophone home monitoring approach to TB was shown to enhance treatment compliance and use less clinic resources in a larger study by Wade et al. (2012).

More recently, Creary et al. (2014) developed a novel mobile DOT approach utilising smartphone and computer devices that resulted in a median monthly observed adherence of 93.3% over the 6 month trial in children with sickle cell disease. Finally, specific to asthma patients, Vasbinder et al., (2013) has developed a study to access the effectiveness of using mobile phone text-messages to remind and encourage non-adherent patients to take their medication and thereby improve control of their disease; results of the study are not yet available. Limited available evidence, therefore, suggests that communication technology could be utilised to achieve therapeutic goals of correct administration technique and improved adherence to therapy in asthma patients while limiting resource utilisation.

The principal aim of this study is to evaluate the feasibility and clinical impact of a mobile DOT approach (via video capture in the patient's home) on the administration technique for, and adherence to, ICS in children with partially controlled or uncontrolled asthma. A secondary aim is to determine factors that influence adherence to ICS in children with asthma.

The specific objectives are to:

1. Investigate the feasibility, practicality, and persistence of a mobile DOT technology approach in the home setting to assist with disease management of children and young people with partially controlled or uncontrolled asthma.
2. Assess inhaler technique and adherence to ICS therapy by use of DOT videos, parent/guardian and child self-report questionnaires (Medication Adherence Report Scale (MARS)), pharmacy records and patient's general practitioner (GP) records.
3. Evaluate the impact of the DOT intervention on asthma clinical outcomes including physician assessment of disease control, medication changes, asthma control tests, health-related quality of life and pulmonary function studies in participating children.
4. Identify parental/guardian and patient factors that influence adherence to ICS in participating children and young people with asthma

ELIGIBILITY:
Inclusion Criteria:

1. Children and young people aged from 2-16 years with apparent partially controlled or uncontrolled DTA. The children will have asthma symptoms despite being prescribed ICS (> 400 mcg/day for children < 5 years, 800 mcg/day for children > 5 years) and a second line therapy such as a LABA, LTRA, or theophylline (Nagakumar and Thomas, 2013).
2. One member of the household has access to a smartphone, tablet or other mobile device that is capable submitting a video image to an internet accessible repository. This person must have access to the device for the entire period of the intervention phase (6 weeks) of the study.

Exclusion Criteria:

1. Children whose asthma symptoms are controlled.
2. Children and/or parents without access or unwilling to allow use of a suitable mobile device for the study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Clinician assessment of asthma control | Recruitment - 18 weeks post intervention
  Clinician assessment of degree of disease control recorded at baseline and during follow-up period
Clinician assessment of asthma severity | Recruitment - 18 weeks post intervention
  Clinician assessment of asthma severity recorded at baseline and during follow-up period
Asthma medication profile | Recruitment - 18 weeks post intervention
  Current medication profile and any changes made
Number of asthma attacks | Recruitment - 18 weeks post intervention
  Number of attacks taken during follow-up period
Oral corticosteroids courses | Recruitment - 18 weeks post intervention
  Numbers of courses of oral corticosteroids taken during follow-up period
Attendances at Emergency Department (ED) | Recruitment - 18 weeks post intervention
  Numbers of attendances to ED during follow-up period
Spirometry measurement; Fraction of exhaled nitric oxide (FeNO) | Recruitment - 18 weeks post intervention
  Measurements taken at each intervention
Self reported Medication Adherence Report Scale (MARS) | Recruitment - 18 weeks post intervention
  Parent/guardian completes MARS if child younger than 9yrs old
Interview-administered Paediatric Asthma Quality of Life Questionnaire (PAQOLQ) or Paediatric Asthma Caregiver Quality of Life Questionnaire (PACQOLQ) | Recruitment - 18 weeks post intervention
  PAQOLQ if 9 years or older; PACQOLQ if under 9
Interview-administered Asthma Control Test (ACT) or Childhood Asthma Control (C-ACT) | Recruitment - 18 weeks post intervention
ICS inhaler technique | Recruitment - 18 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mike Shields, PhD, Principal Investigator — Queen's University, Belfast